CLINICAL TRIAL: NCT05557422
Title: Clinical Performance Evaluation of the BD OneFlow CLPD Panel (BD OneFlow LST, and B-CLPD T1 to T4 Assays) on the BD FACSLyric System.
Brief Title: BD OneFlow CLPD Panel (BD OneFlow LST, and B-CLPD T1 to T4 Assays) on the BD FACSLyric System.
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CAS-OFLBT1T4
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-03

CONDITIONS: Chronic Lymphoproliferative Diseases (CLPD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: BD OneFlow LST, and B-CLPD T1 to T4 Assays — a panel of fluorochrome-conjugated antibodies for qualitative flow-cytometric immunophenotyping of mature lymphocyte populations on the BD FACSLyric™ flow cytometer with BD FACSuite™ Clinical application.

SUMMARY:
Multi-site, prospective performance study to determine equivalency between the investigational CLPD Full Panel on the FACSLyric system versus the final clinical diagnosis.

DETAILED DESCRIPTION:
This study is a multi-site and multi-regional prospective performance evaluation to determine sensitivity and specificity of the investigational BD OneFlow CLPD Panel on the FACSLyric system when compared to the results from the Expert Analysis for market launch.

The study will be conducted at up to eight investigational sites that have previously participated in the BD OneFlow program clinical studies and/or have expertise in flow cytometric immunophenotyping, interpretation, and diagnosis of Leukemia and Lymphoma (L&L). Each site will have one 10- or 12-color FACSLyric instrument with Universal Loader (Loader).

This study will enroll at least 250 leftover de-identified PB, BM, and LT specimens from routine flow cytometry laboratory testing for hematological disorders or non-hematological disorders that provide valid results and are considered evaluable specimens. Each site will enroll a minimum of 25 evaluable specimens and a maximum of approximately 70 evaluable specimens with normal and abnormal lymphoid cell immunophenotype.

To ensure that the study satisfies enrollment by specimen type, this study will enroll lymphoid tissue specimens. Lymphoid tissue (LT) refers to organs/tissues supporting immune responses, which includes primary lymphoid tissue (BM and thymus), and secondary lymphoid tissue (lymph nodes, tonsils, spleen, and Peyer's patches). Their morphological structure is related to its function in the immune system. For this study, the term LT will be used to refer the secondary lymphoid tissue only.

Evaluable specimens will be enrolled to meet the binning requirements for specimen type, normal vs abnormal cell phenotype, and disease type, as described in Tables 3-5.

Specimens will be prepared using a minimum of three lots of the OneFlow LST and OneFlow B-CLPD T1 to T4 reagent kits across investigational sites. Stained samples will be acquired on the BD FACSLyric using the BD FACSuite Clinical application with the assay modules for each of the tubes. Results will be analyzed by the laboratory staff. In addition, the sites will collect the "Final Clinical Diagnosis" from each sample.

The study includes an "Expert Analysis." This will be conducted by qualified Experts by training and experience, who will receive the files with raw data, analyze and designate cell immune phenotype. Two Experts will analyze the data from each sample. The results from the Expert Analysis will be compared to the site's Final Clinical Diagnosis and the study acceptance criteria for the study endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Specimen collected/handled prior to enrollment in accordance with site policies and procedures.
2. Specimen with adequate volume (min 700 µL or more) to complete protocol tests.
3. Specimen is leftover PB, BM, or LT from routine flow cytometry laboratory testing for chronic lymphoproliferative disorders, other hematological disorders, non-hematological tumors (e.g., solid tumors), or other hematological disorders (non-malignant).
4. Specimen is from subjects previous diagnosed, newly diagnosed and/or relapsed disease.
5. Only one type of specimen, either PB, BM, or LT shall be enrolled per given subject.
6. Specimen is stored at room temperature, upon receipt by the site.
7. PB and BM specimens are collected in EDTA (K2 or K3) or heparin (sodium or lithium).
8. LT specimens collected in PBS, culture media (e.g., RPMI-1640), saline, or saline wrapped gauze at the discretion of the Investigator.
9. Age of specimen for PB and BM (time of collection to start of first pre-wash): ≤ 24 hours. (Note: No Age of specimen claim is being made for LT)
10. Specimens are from subjects irrespective of race, gender, and ethnicity

Exclusion Criteria:

1. Specimen is from healthy subject.
2. Specimen is from subject undergoing any treatment for any form of L&L.
3. Specimen from subject <22 years of age.
4. Specimen is from subject with minimal residual disease (MRD) as determined by the site.
5. Specimen is from subject suspected of acute leukemia (e.g., T-ALL, BCP-ALL, AML) or myeloid dysplastic syndrome (MDS).
6. Visibly clotted specimen.
7. Visibly hemolyzed specimen.
8. Frozen specimen.
9. Refrigerated specimen.
10. Fixed specimen.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of evaluable 250 remnant/leftover peripheral blood, bone marrow, and lymph node specimens from routine flow cytometry laboratory testing for hematological disorders. Specimens from healthy subjects will be excluded.
  Specimens are from subjects irrespective of race, gender, and ethnicity. Specimen from subject >22 years of age .
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Comparison between expert analysis determination for normal and abnormal specimen and final dignosis | Age of Specimen for PB and BM (time of collection to start of first pre-washed) <24 hours
  Determine equivalence between the investigational OneFlow CLPD panel on FACSLyric system results analyzed by two independent experts versus the final clinical diagnosis for Normal (T-cell, B-cell, and NK-cell) or Abnormal (T-cell or B-cell or NK-cell) phenotype using leftover, hematologically abnormal specimens.

SECONDARY OUTCOMES:
Comparison between expert analysis determination for normal and abnormal Peripheral Blood (PB) specimen and final dignosis | ge of Specimen for PB (time of collection to start of first pre-washed) <24 hours.
  Supplement equivalence between the investigational OneFlow CLPD on FACSLyric system results analyzed by two independent experts versus the final clinical diagnosis for Normal (T-cell, B-cell, and NK-cell) or Abnormal (T-cell or B-cell or NK-cell) phenotype using leftover, hematologically abnormal peripheral blood (PB) specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Imelda Omana-Zapata, MD, Ph.D, Study Director — Becton, Dickinson and Company
Locations (6):
- United States (2):
  - University of Norht Calolina, Chapel Hill, North Carolina
  - CorePATH Laboratories, San Antonio, Texas
- Erasmus Medical Center, Laboratory Medical Immunology, Department of Immunology, Rotterdam, Netherlands
- Champalimaud Foundation, Lisbon, Portugal
- University of Salamanca, Salamanca, Spain
- Kantonsspital Aarau AG / IfLM, Aarau, Switzerland

IPD SHARING:
Plan to Share IPD: No